CLINICAL TRIAL: NCT00183703
Title: Rapid Cycling Bipolar Disorder (RCBPD), Subjective Illness Experience and Gender
Brief Title: Understanding Treatment Adherence Among Individuals With Rapid Cycling Bipolar Disorder
Status: Completed | Type: Observational
Sponsor: Case Western Reserve University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Martha Sajatovic, MD, Professor of Psychiatry and of Neurology, Case Western Reserve University
Other Study IDs: K23MH065599-02 (NIH); K23MH065599-02 (NIH)
Record Dates: First submitted 2005-09-14; First posted 2005-09-16 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Bipolar Disorder
Keywords: Depression, Bipolar; Manic-Depressive Psychosis
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Qualitative Interview: Participants with rapid cycling bipolar disorder (RCBPD)

SUMMARY:
This study will examine how various factors, such as psychiatric symptoms, gender, quality of life, and attitudes toward medication, affect treatment adherence in individuals with rapid cycling bipolar disorder.

DETAILED DESCRIPTION:
Bipolar Disorder (BPD), also known as manic-depressive illness, is a disorder that causes frequent shifts in an individual's mood, energy, and ability to function. An individual with BPD may go through periods of mania, which are characterized by increased energy, irritability, and an excessively "high" euphoric mood. The manic periods are followed by periods of depression, which are characterized by decreased energy, feelings of hopelessness, and anxiety. Rapid cycling bipolar disorder (RCBPD) is a type of BPD in which the individual experiences four or more episodes of mania and depression per year. The rapid shift between the manic and depressive episodes makes it imperative that individuals with RCBPD strictly manage their illness with medication. Many BPD medications have been developed recently; however, there are still many individuals who do not respond well to medication treatment. Research has shown that the way individuals experience illness has an effect on their response to medication. The purpose of this study is to gain insight into how individuals with RCBPD perceive and respond to medication treatment. Factors such as gender, degree of social support, drug and alcohol usage, and attitudes towards medication will be evaluated to understand how they affect medication and treatment adherence.

This study will consist of 1 visit, which will last approximately 2 and ½ hours and will include an anthropological interview and numerous standardized psychological questionnaires. The interview and questionnaires will assess participants' attitudes toward BPD treatment; psychiatric illness severity, including symptoms of mania and depression; expectations regarding recovery, stigma, and quality of life; and medication adherence.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of rapid cycling variant of bipolar disorder type I; diagnosed 2 to 20 years prior to study entry
* Has experienced an index depressive episode
* Received treatment with medication to stabilize mood for at least 6 months prior to study entry
* Lives in the Northeast Ohio area and is a patient at either Northeast Ohio Health Services or The Mood Disorders Clinic at University Hospitals of Cleveland

Exclusion Criteria:

* Unable/unwilling to participate in psychiatric interviews

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population includes 20 individuals receiving treatment at an academic medical center and 20 individuals seeking treatment at a community mental health clinic.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2004-07; Primary Completion 2006-11 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
The Subjective Experience of Medication Interview (SEMI) | Baseline
  The Subjective Experience of Medication Interview (SEMI) is a qualitative, semi-structured assessment of subjective experience of mental illness, which requires approximately 60-120 minutes to administer. Illness experience domains assessed include illness attitudes, attributions and behaviors, social relations, treatment history and medication experience, self-medication, quality of life, stigma, culture/ethnicity, and health care logistics. The SEMI has been modified for use in populations with Bipolar Disorder.

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale (HAMD) | Baseline
  A rater administered rating to scale to measure symptoms of depression, and is the most commonly utilized rating scale to assess depressive symptoms in bipolar depression clinical studies.
Clinical Global Impression (CGI) | Baseline
  Global illness severity is measured with the Clinical Global Impressions (CGI), a widely used scale which evaluates illness severity on a 1 to 7 point continuum. Severity of illness ratings on the CGI have reported reliability scores ranging from 0.66-0.41.
Insight and Treatment Attitudes Questionnaire (ITAQ) | Baseline
  An 11-item rating scale to evaluate patient recognition of illness and need for treatment in psychiatric illness. Each ITAQ item is scored on a 0 to 2 scale (0 = no insight, 2 = good insight), and the scale has high interrater reliability (r=0.82, p<.001) (McEvoy 1981). Construct validity, checked by correlating scores with an open interview is also good (r=.85, p<.001).
Illness Behavior Questionnaire (IBQ) | Baseline
  A 62-item instrument designed to measure a respondent's attitudes, ideas, affects and attributions in relation to illness. The IBQ is a self-reported scale, in which the respondent answers "yes" or "no" to each question regarding illness experience and subjective response. There are seven major subscales derived through factor analysis. The IBQ has very good stability, with one-to-twelve week test-retest correlations ranging from .67-.85 for the subscales. It has good face and content validity.
Attitude Towards Mood Stabilizers Questionnaire (AMSQ) | Baseline
  A modification of the Lithium Attitudes Questionnaire (Harvey 1991) which evaluates an individual's attitudes towards mood stabilizing medication (Adams and Scott 2000). The AMSQ comprises 19 items grouped into 7 subscales: general opposition to prophylaxis (4 items), denial of illness severity (3 items), negative attitudes toward drugs in general (3 items), and lack of information about mood stabilizers (1 item). Higher scores on each subscale represent more negative attitudes toward mood stabilizers. Reliability for the 19 items ranges from 57.6 % to 96.9%.
Multidimensional Health Locus of Control Scale (MHLC) | Baseline
  An 18-item instrument that measures three dimensions of locus of control of reinforcement as it pertains to health (internal, IHLC: external-chance, CHLC: and external powerful others, PHLC). Scoring is from 6-36 with higher scores indicating stronger beliefs. The internal consistency reliability using Cronbach's alpha ranges from .67 to .77 for the three dimensions, and the measure has fairly good criterion validity (Wallston 1978).
Treatment Adherence | Baseline
  Treatment adherence will be evaluated in the following three ways: 1) The primary measure will be the Tablet Routines Questionnaire (TRQ, Peet 1991) which is a validated assessment of adherence among individuals with bipolar disorders (Scott 2002, Peet 1991), 2) Blood level of mood stabilizing and antipsychotic medications will be identified from the patient record. This has been identified as a standard of care in numerous guidelines for the treatment of bipolar disorder (American Psychiatric Association 2000, Goldberg 2000). 3) Adherence with clinic visits for the previous three month time period will be calculated as a percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Martha Sajatovic, MD, Principal Investigator — Case Western Reserve University School of Medicine
Locations (2):
- United States (2):
  - Northeast Ohio Health Services, Beachwood, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio

REFERENCES:
- [Result] Sajatovic M, Jenkins JH, Cassidy KA, Muzina DJ. Medication treatment perceptions, concerns and expectations among depressed individuals with Type I Bipolar Disorder. J Affect Disord. 2009 Jun;115(3):360-6. doi: 10.1016/j.jad.2008.10.002. Epub 2008 Nov 8. PMID 18996600
- [Result] Sajatovic M, Jenkins JH, Safavi R, West JA, Cassidy KA, Meyer WJ, Calabrese JR. Personal and societal construction of illness among individuals with rapid-cycling bipolar disorder: a life-trajectory perspective. Am J Geriatr Psychiatry. 2008 Sep;16(9):718-26. doi: 10.1097/JGP.0b013e3180488346. Epub 2007 Dec 10. PMID 18070834